CLINICAL TRIAL: NCT00320359
Title: An Open-Label, Multicentre, Randomised, Phase III Study Comparing Topotecan/Cisplatin and Topotecan/Etoposide Versus Etoposide/Cisplatin as Treatment for Chemotherapy-naive Patients With Extensive Disease-Small Cell Lung Cancer
Brief Title: Topotecan Plus Cisplatin Versus Etoposide Plus Cisplatin In 1st Line Extensive Disease Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104864-A/479
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Lung Cancer, Small Cell
Keywords: First-line Cisplatin; Small Cell Lung Cancer; topotecan; etoposide; Extensive Disease
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Cisplatin

ARMS (2):
- Arm A (Active Comparator): Cisplatin 75 mg/m2 i.v., day 1, Etoposide 100 mg/m2 i.v., days 1-3
  Interventions: Drug: Intravenous etoposide/cisplatin
- Arm B (Experimental): Topotecan 1 mg/ m2, i.v., days 1-5 Cisplatin 75 mg/m2 i.v., days 5
  Interventions: Drug: Intravenous topotecan/cisplatin

INTERVENTIONS:
Drug: Intravenous topotecan/cisplatin — Topotecan 1 mg/m2 should be administered intravenously over a period of 30 minutes on days 1-5. Then a 30 minute saline flush should be administered followed by the cisplatin on day 5.
  Cisplatin 75 mg/m2 given as an intravenous infusion at the rate of 1 mg/min on day 5 after topotecan.
  Arms: Arm B
Drug: Intravenous etoposide/cisplatin — Cisplatin 75 mg/m2 given as an intravenous infusion at the rate of 1 mg/min on day 1. Cisplatin should be given simultaneously to post-hydration to ensure a high volume fluid.
  Etoposide 100 mg/m2 should be administered after cisplatin intravenously over a period not less than 30 minutes on days 1 -3.
  Arms: Arm A

SUMMARY:
Evaluation of intravenous Topotecan + Cisplatin as a potential new standard of care in 1st line Small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

* Evaluable extensive small cell lung cancer, extensive disease.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2.
* Life expectancy > 3 months.
* Fit to receive any of the treatments.
* No prior chemotherapy.
* Written informed consent.

Exclusion Criteria:

* Extensive disease treatable with radiotherapy.
* Past or current history of other malignant disease.
* Prior chemotherapy.
* Pregnancy, lactating or lack of effective contraception.
* Concurrent severe medical problems other than small cell lung cancer.
* Patients with central nervous system metastases receiving more than 12 mg /day dexamethasone or equivalent to control symptoms.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2002-08; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Median overall survival time of participants | Up to 1 year after randomization of the last patient

SECONDARY OUTCOMES:
Number of participants with one year survival rate of the participants | Up to 1 year after randomization of the last patient
Median time of disease progression | up to 1 year after randomization of the last patient
Median time to event (progressive disease or death) of participants | Up to 1 year after randomization of the last patient
Median time to response to chemotherapy | Up to 1 year after randomization of the last patient
Median response duration | Up to 1 year after randomization of the last patient
Number of participants with objective response | Up to 1 year after randomization of the last patient
Mean lung cancer symptom score (LCSS) | Up to 18 weeks
Mean eastern cooperative oncology group (ECOG) score | Up to 18 weeks
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to 1 year after randomization of the last patient
Mean change from Baseline in hemoglobin value | Baseline and up to 18 weeks
Mean change from Baseline in leukocytes, neutrophils and platelets count | Baseline and up to 18 weeks
Mean change from Baseline in red blood cells (RBCs) | Baseline and up to 18 weeks
Mean change from Baseline in Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alkaline phosphatase and Lactate dehydrogenase (LDH) | Baseline and up to 18 weeks
Mean change from Baseline in Blood urea nitrogen (BUN), Potassium, Sodium and urea | Baseline and up to 18 weeks
Mean change from Baseline in Creatinine and Total bilirubin | Baseline and up to 18 weeks
Mean change from Baseline in Creatinine clearance
Mean change from Baseline in total protein | Baseline and up to 18 weeks
Number of participants with abnormal urinalysis results
Mean change from Baseline in weight | Baseline and up to 18 weeks
Mean change from Baseline in Body surface area | Baseline and up to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (64):
- Austria (4):
  - GSK Investigational Site, Bludesch
  - GSK Investigational Site, Klagenfurt
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Vienna
- Germany (60):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Löwenstein, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Wangen, Baden-Wurttemberg
  - GSK Investigational Site, Bayreuth, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Passau, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Rosenheim, Bavaria
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Frankfurt (Oder), Brandenburg
  - GSK Investigational Site, Bremen, City state Bremen
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Giessen, Hesse
  - GSK Investigational Site, Greifenstein, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Limburg an der Lahn, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Offenbach, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Leer, Lower Saxony
  - GSK Investigational Site, Stade, Lower Saxony
  - GSK Investigational Site, Greifswald, Mecklenburg-Vorpommern
  - GSK Investigational Site, Neubrandenburg, Mecklenburg-Vorpommern
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Stralsund, Mecklenburg-Vorpommern
  - GSK Investigational Site, Waren, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Coesfeld, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dorsten, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Hamm, North Rhine-Westphalia
  - GSK Investigational Site, Hemer, North Rhine-Westphalia
  - GSK Investigational Site, Herne, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Oberhausen, North Rhine-Westphalia
  - GSK Investigational Site, Velbert, North Rhine-Westphalia
  - GSK Investigational Site, Wuppertal, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Plauen, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Borstel, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Erfurt, Thuringia
  - GSK Investigational Site, Jena, Thuringia